CLINICAL TRIAL: NCT01323218
Title: Effect of the Correction of Vitamin D Deficiency in Patients With Obstructive Sleep Apnea-hypopopnea Syndrome (OSAHS)
Brief Title: Sleep Apnea Syndrome and Vitamin D
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Recherche en Nutrition Humaine d'Auvergne (Other Government); Centre de Recherche en Nutrition Humaine Rhone-Alpe (Other); Laboratoire Crinex (Unknown); Laboratoire Cidelec (Unknown)
Responsible Party: Patrick LACARIN, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0091
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2011-03-25 (Estimated); Status verified 2011-03

CONDITIONS: Obstructive Sleep Apnea-hypopnea Syndrome
Keywords: Obstructive sleep apnea-hypopnea syndrome; OSAHS; Vitamin D
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: 25 OH vitamin D — After written informed consent, patients will be randomized to receive a single dose of oral vitamin D (400 000 UI) or placebo. Subjects will undergo medical screening before randomisation into placebo or active group. Follow-up measurements will be performed at the beginning (day 0) and after 32 days of vitamin D supplementation: clinical examination, biological check up and sleep parameter evaluation. Patients will be instructed to stop using continuous positive airway pressure device for two nights before nocturnal sleep studies

SUMMARY:
Obstructive sleep apnea/hypopnea syndrome (OSAHS) is a highly prevalent disorder with multiple comorbidities.

OSAHS is characterized by repetitive episodes of airflow reduction (hypopnoea) or cessation (apnoea) due to upper airway collapse during sleep. Its major risk factor is obesity. However, its pathogenesis is complex and multifactorial. Reduced upper airway muscle tonus and/or unstable neuromuscular output seem to be involved in this collapsus.

A normal vitamin D status is necessary for normal muscle function and neuromuscular output. As obesity is associated with a high rate of hypovitaminosis D, it appears of interest to evaluate the effect of vitamin D supplementation on OSAHS patients with vitamin D deficiency.

DETAILED DESCRIPTION:
Prospective, longitudinal, double bind, randomized study of the effect of vitamin D supplementation in OSAHS patients with hypovitaminosis D.

After written informed consent, patients will be randomized to receive a single dose of oral vitamin D (400 000 UI) or placebo. Subjects will undergo medical screening before randomisation into placebo or active group. Follow-up measurements will be performed at the beginning (day 0) and after 32 days of vitamin D supplementation: clinical examination, biological check up and sleep parameter evaluation. Patients will be instructed to stop using continuous positive airway pressure device for two nights before nocturnal sleep studies.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe obstructive sleep apnoea (AHI > 15)
* With or without continuous positive airway pressure for a minimum of six months
* aged 30-75 years
* Vitamin D2D3 level < 30 ng/ml

Exclusion Criteria:

* Diseases or therapy known to interfere with phospho-calcium or vitamin D metabolism
* Patients with mixed sleep apnoea (central and obstructive)
* Patients with CPAP use < 4 hours per night
* Patients with maxillofacial or oro-pharyngeal diseases)
* Patients with chronic respiratory failure, hypercapnic patients
* Muscle diseases
* Alcohol intake > 2 glasses per day
* Body mass index > 40 kg/m2

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-04 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI), defined as the average rate of apneas and hypopneas per hour of sleep | at the beginning (day 0) and after 32 days of vitamin D supplementation

SECONDARY OUTCOMES:
Epworth sleepiness scale | at the beginning (day 0) and after 32 days of vitamin D supplementation
mean arterial oxygen saturation (SaO2) during sleep, time of SaO2<90%, and Nadir of arterial oxygen saturation (Nadir SaO2) | at the beginning (day 0) and after 32 days of vitamin D supplementation
Continuous positive airway pressure measured with a CPAP equipment | at the beginning (day 0) and after 32 days of vitamin D supplementation
Muscular strength measured with handgrip test | at the beginning (day 0) and after 32 days of vitamin D supplementation
Mini Mental Sate Examination, trail making test, Hamilton Anxiety Depression scale, SF36 questionnaire | at the beginning (day 0) and after 32 days of vitamin D supplementation
Inflammatory status : IL6 and high sensitivity C-reactive proteine (hs CRP) | at the beginning (day 0) and after 32 days of vitamin D supplementation
Analysis of genes implicated in vitamin D metabolism | at inclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France